CLINICAL TRIAL: NCT06111014
Title: A Continuation Study of Latozinemab in Participants With Neurodegenerative Disease
Brief Title: Continuation Study for Latozinemab
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The AL001-CS-302 study was terminated because its Phase 3 placebo-controlled parent study (AL001-3) failed to meet the clinical co-primary endpoint of slowing FTD-GRN progression, as measured by the Clinical Dementia Rating® plus National Alzheimer's
Sponsor: Alector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL001-CS-302; 2023-506805-20-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-10-18; First posted 2023-11-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neurodegenerative Diseases
Keywords: Frontotemporal Dementia (FTD); Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Neurodegenerative Diseases; Frontotemporal Dementia; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Open-label
Masking Description: This is an open label continuation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Latozinemab (AL001) administered by IV infusion over 60 minutes, q4w
  Interventions: Drug: Latozinemab

INTERVENTIONS:
Drug: Latozinemab — All participants will receive open-label latozinemab at a dose of 60/mg/kg, every 4 weeks
  Other Names: AL001

SUMMARY:
Continuation study to provide continued access to latozinemab for participants who have previously participated in a latozinemab study

DETAILED DESCRIPTION:
This is an open-label continuation study to provide access and assess the safety and tolerability of latozinemab in participants who have completed participation in their parent latozinemab study.

All participants will receive open-label latozinemab at a dose of 60/mg/kg, every 4 weeks (q4w).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented (from the participant or, where jurisdictions allow it, from their legal decision maker).
* Has successfully completed participation in their parent latozinemab study.
* Female participants must be nonpregnant and nonlactating.
* Male participants must agree to acceptable contraception use.

Exclusion Criteria:

* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins.
* Clinically significant heart disease, liver disease or kidney disease. History or evidence of clinically significant brain disease other than FTD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Number of participants receiving latozinemab | Through study completion, up to 190 weeks
  Number of participants receiving latozinemab
Duration of treatment with latozinemab | Through study completion, up to 190 weeks
  Duration of treatment with latozinemab

SECONDARY OUTCOMES:
Incident of adverse events (AEs) and serious adverse events (SAEs) | Through study completion, up to 190 weeks
  Number and percentage of participants of AEs or SAEs
Nature and severity of AEs and SAEs | Through study completion, up to 190 weeks
  Severity of AEs and SAEs according to the World Health Organization (WHO) toxicity grading scale
Incidence of ADAs to latozinemab | Through study completion, up to 190 weeks
  Number and percentage of participants with anti-Drug Antibodies (ADA) titer over study time points

CONTACTS AND LOCATIONS:
Overall Officials: Study Lead, Study Director — Alector Inc.
Locations (18):
- United States (5):
  - Dignity Health - Arizona, Phoenix, Arizona
  - Mayo Comprehensive Cancer Center - PPDS, Rochester, Minnesota
  - Irving Institute for Clinical and Translational Research, New York, New York
  - University of Cincinnati Gardner Neuroscience Institute, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - Parkwood Institute, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Groupe Hospitalier Pitié Salpétrière, Paris, France
- Universitätsklinikum Ulm - Leimgrubenweg 12-14, Ulm, Germany
- Italy (3):
  - IRCCS - Centro S. Giovanni di Dio Fatebenefratelli, Brescia
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico -Via Fracesco Sforza 35, Milan
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena
- Erasmus MC-Dr. Molewaterplein 40, Rotterdam, Netherlands
- Portugal (2):
  - Centro Hospitalar E Universitario de Coimbra EPE, Coimbra
  - Centro Hospitalar Universitário Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
- Karolinska Universitetssjukhuset Huddinge, Huddinge, Sweden
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No